CLINICAL TRIAL: NCT00644488
Title: A Phase I Study of BMS-641988 in Japanese Patients With Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA185-005
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2009-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BMS 641988

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A1 (Experimental): Active
  Interventions: Drug: BMS-641988 (AR#2)

INTERVENTIONS:
Drug: BMS-641988 (AR#2) — Tablets, Oral, 20 mg, 40 mg, 60 mg, 100 mg, once daily, 24 weeks

SUMMARY:
The purpose of this clinical study is to assess the safety and tolerability of BMS-641988 once daily orally in Japanese patients with castration resistant prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with castration-resistant prostate cancer and serum testosterone ≤50 ng/dL progressive to current therapy who satisfy the inclusion and exclusion criteria

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of BMS-641988 once daily orally in Japanese patients with castration resistant prostate cancer | throughout the study

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of BMS-641988 and the metabolites BMS-501949 and BMS-570511 | at cycle 1 day 1, day 15 and day 29
To identify the dose(s) of BMS-641988 for Phase II | at the end of study
To assess any preliminary evidence of anti-tumor activity by PSA decline, tumor shrinkage, radionuclide bone scans | throughout the study
To assess the effects of BMS-641988 on pharmacodynamic markers (LH, total and free testosterone, 5(alpha)-DHT, estradiol, prolactin, FSH, and SHBG) | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Japan (3):
  - Local Institution, Hidaka, Saitama
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Koto-Ku, Tokyo

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx